CLINICAL TRIAL: NCT02969681
Title: A Randomized Phase Ⅲ Study of IV Ascorbic Acid in Combination With FOLFOX+/- Bevacizumab vs Treatment With FOLFOX+/- Bevacizumab Alone as First-line Therapy for Advanced Colorectal Cancer
Brief Title: Vitamin C Intravenously With Chemotherapy in Advanced Colorectal Cancer
Acronym: Vitality
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VitC001
Record Dates: First submitted 2016-05-15; First posted 2016-11-21 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ascorbic Acid; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ascorbic Acid with chemotherapy group (Experimental): Ascorbic Acid with mFOLFOX6 with or without bevacizumab Ascorbic Acid (1.5g/kg/day, D1-3) every 2 weeks
  mFOLFOX6:
  * Oxaliplatin 85 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  with or without bevacizumab 5mg/kg, every 2 weeks
  Interventions: Drug: ascorbic acid; Drug: Chemotherapy
- Chemotherapy group (Active Comparator): mFOLFOX6:
  * Oxaliplatin 85 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  with or without bevacizumab 5mg/kg, every 2 weeks
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: ascorbic acid — 1.5g/kg/day, D1-3, every 2 weeks
  Other Names: Vitamin C
  Arms: Ascorbic Acid with chemotherapy group
Drug: Chemotherapy — * mFOLFOX6
  * Oxaliplatin 85 mg/m² d1 concurrent with
  * Leucovorin 400 mg/m², followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 2400 mg/m² over 46 hours, every 2 weeks
  with or without bevacizumab 5mg/kg, every 2 weeks
  Other Names: mFOLFOX6+/- bevacizumab

SUMMARY:
Preclinical study has shown that human colorectal cancer cells harboring KRAS or BRAF mutations are selectively killed by high levels of ascorbic acid (AA). High dose of AA aslo impairs tumor growth in Apc/KRASG12D mutant mice. Previous phase Ⅰ studies have found that high dose iv AA is well tolerated in cancer patients.This protocol is a phase Ⅲ study of AA infusions combined with treatment with FOLFOX +/- bevacizumab versus treatment with FOLFOX +/- bevacizumab alone as first-line therapy in patients with recurrent or advanced colorectal cancer.

DETAILED DESCRIPTION:
Linus Pauling and Dr Ewan Cameron have published two retrospective studies about using high dose vitamin C to treat cancer patients forty years ago. Their studies have shown that high dose vitamin C usage could significantly prolong overall survival of patients with advanced cancer. Recently, preclinical study has shown that human colorectal cancer cells harboring KRAS or BRAF mutations are selectively killed by high levels of ascorbic acid (AA). High dose of AA impairs tumor growth in Apc/KRASG12D mutant mice. Previous phaseⅠ clinical trials have found that high dose (1.5g/kg or 90g/m2) iv AA is well tolerated in cancer patients. This protocol is a phase Ⅲ, study of ascorbic acid (AA) infusions combined with treatment with FOLFOX +/- bevacizumab versus treatment with FOLFOX +/- bevacizumab alone as first-line therapy in patients with recurrent or advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Age≥18 years, ≤75 years; Histologically proven metastatic adenocarcinoma of colorectal cancer (stage Ⅳ disease), unresectable metastatic disease; measurable disease; G6PD status > lower limit of normal; Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1; Life expectancy of at least 12 weeks; ANC ≥1,500/mm3; Hemoglobin > 8g/dL; platelet ≥ 100,000/mm3; Laboratory at baseline evaluation for inclusion in the study: creatinine ≤1.5X upper limit [if the creatinine is elevated, but ≤1.5X the ULN, a 24 hour creatinine clearance will be obtained, Creatinine clearance > 50 mL/min (calculated according to Cockroft and Gault)]; Transaminase (AST/ALT) ≤2.5X upper limit of normal and bilirubin levels ≤1.5X upper limit of normal without liver metastasis; Transaminase (AST/ALT) ≤5X upper limit of normal and bilirubin levels ≤1.5X upper limit of normal with liver metastasis; Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the study; Written informed consent

Exclusion Criteria:

Prior treatment for metastatic disease (adjuvant therapy with fluoropyrimidines +/-oxaliplatin based regimens allowed if stopped 12 months prior to registration on study); Surgery (excluding diagnostic biopsy) or irradiation within 3 weeks prior to study entry; Administration of any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment; Concurrent chronic systemic immune therapy, chemotherapy, radiation therapy (palliative radiation therapy allowed) or hormone therapy not indicated in the study protocol; Brain metastasis (known or suspected); Pregnant or lactating women; Other uncontrolled concomitant illness, including serious uncontrolled intercurrent infection; Known allergy or any other adverse reaction to any of the drugs or to any related compound; Previous (within 5 years) or concurrent malignancies at other sites with the exception of surgically cured or adequately treated carcinoma in-situ of the cervix and basal cell carcinoma of the skin; Patients who are on strong inducers of CYP3A4 which include but are not limited to: Aminoglutethimide, Bexarotene, Bosentan, Carbamazepine, Dexamethasone, Efavirenz, Fosphenytoin, Griseofulvin, Modafinil, Nafcillin, Nevirapine, Oxcarbazepine, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, Rifapentine, St. John's wort; Medical, social or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent; Organ allograft requiring immunosuppressive therapy; Patients with HIV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2017-01; Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | up to 5 years
  Time-to-event outcome measure (initial disease progression) measured in days from cycle 1 day 1 to day of first progression as defined by RECIST1.1 criteria from NCI

SECONDARY OUTCOMES:
Overall Survival | up to 5 years
  Time to event outcome measure (death), measured in days from cycle 1 day 1
Response Rate | up to 5 years
  To utilize CT or PET/CT scans to assess overall tumor response rate (complete and partial response) and evaluate disease progression in subjects with advanced or recurrent RAS mutant colorectal cancer treated with the combination of ascorbic acid and FOLOX/FORFIRI +/- bevacizumab versus treatment with FOLFOX/FORFIRI +/- bevacizumab alone
Assessment of treatment-related adverse events | up to 5 years
  Assessment of the percentage of participants with adverse events and serious adverse events observed throughout the study, and for 30 days after cessation of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD.,PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yun J, Mullarky E, Lu C, Bosch KN, Kavalier A, Rivera K, Roper J, Chio II, Giannopoulou EG, Rago C, Muley A, Asara JM, Paik J, Elemento O, Chen Z, Pappin DJ, Dow LE, Papadopoulos N, Gross SS, Cantley LC. Vitamin C selectively kills KRAS and BRAF mutant colorectal cancer cells by targeting GAPDH. Science. 2015 Dec 11;350(6266):1391-6. doi: 10.1126/science.aaa5004. Epub 2015 Nov 5. PMID 26541605
- [Background] Hoffer LJ, Levine M, Assouline S, Melnychuk D, Padayatty SJ, Rosadiuk K, Rousseau C, Robitaille L, Miller WH Jr. Phase I clinical trial of i.v. ascorbic acid in advanced malignancy. Ann Oncol. 2008 Nov;19(11):1969-74. doi: 10.1093/annonc/mdn377. Epub 2008 Jun 9. PMID 18544557
- [Background] Stephenson CM, Levin RD, Spector T, Lis CG. Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetics of high-dose intravenous ascorbic acid in patients with advanced cancer. Cancer Chemother Pharmacol. 2013 Jul;72(1):139-46. doi: 10.1007/s00280-013-2179-9. Epub 2013 May 14. PMID 23670640
- [Derived] Wang F, He MM, Wang ZX, Li S, Jin Y, Ren C, Shi SM, Bi BT, Chen SZ, Lv ZD, Hu JJ, Wang ZQ, Wang FH, Wang DS, Li YH, Xu RH. Phase I study of high-dose ascorbic acid with mFOLFOX6 or FOLFIRI in patients with metastatic colorectal cancer or gastric cancer. BMC Cancer. 2019 May 16;19(1):460. doi: 10.1186/s12885-019-5696-z. PMID 31096937